CLINICAL TRIAL: NCT04820920
Title: Online Learning Through Play Plus Culturally Adapted Cognitive Behaviour Therapy (LTP+CaCBT) for Treating Depression in British Mothers of African and Caribbean Heritage: A Pilot Randomised Controlled Trial
Brief Title: Online LTP+CaCBT for Treating Depression in British Mothers of African/Caribbean Heritage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nottingham Trent University (Other)
Collaborators: University of Manchester (Other); Teesside University (Other); Sheffield Hallam University (Other)
Responsible Party: Principal Investigator, Dr Dung Jidong, PhD, Senior Lecturer, Nottingham Trent University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0000-0001-5034-0335a
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Postnatal Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LTP+CaCBT (Experimental): The LTP+CaCBT intervention will consist of 10 (mother-child pairs) participants per sub-group in online group sessions (approx. 60 minutes each) and will deliver one session every fortnight for 12 sessions.
  Interventions: Behavioral: LTP; Behavioral: CaCBT
- Psychoeducation (Active Comparator): This is a form of psychoeducation involving basic discussions around mother-child relationships, childcare, child nursing related activities and general maternal discussions. The psychoeducation would last approximately 60 minutes each for 12 sessions (10 participants per sub-group). One session would be delivered every fortnight for 12 sessions.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: LTP — LTP is a low-literacy, sustainable programme that will provide depressed mothers with valuable skills on parenting, improve mother-child relation and mental health self-care. This is a research-based activity that enhances postnatal mental health while simultaneously promoting attachment security through building parents' ability to monitor and be sensitive to their children's cues, and thereby, actively involves in their children's mental and physical development.
  Other Names: Learning Through Play
  Arms: LTP+CaCBT
Behavioral: CaCBT — CaCBT adopts 'here and now' problem-solving approach, which involves collaborating with families, active listening techniques, changing negative thinking, and depressive symptoms associated with postnatal depression and other forms of parenting distress.
  Other Names: Cultural adapted Cognitive and Behaviour Therapy
  Arms: LTP+CaCBT
Behavioral: Psychoeducation — This is a form of psychoeducation involving basic discussions around mother-child relationships, childcare, child nursing related activities and general maternal discussions.
  Arms: Psychoeducation

SUMMARY:
The pilot trial aims to test the feasibility, acceptability and cultural appropriateness of online LTP+CaCBT for treating postnatal depression and to improve the mental health and wellbeing of mothers and their children in the UK.

DETAILED DESCRIPTION:
Participants who scored 5 or above on Patient Health Questionnaire (PHQ-9) will be would be recruited and randomly assigned into one of two groups (experimental or controlled). Experimental groups will receive the online LTP+CaCBT treatment - the intervention will consist of a total of 12 group training sessions (approx. 60 minutes each). The controlled groups will receive 'placebo effects' in the form of psychoeducation involving basic discussions around mother-child relationships, childcare, child nursing related activities and general maternal discussions. Each of the two groups (both experimental and controlled) will be comprised of approximately 10 mother-child pairs per sub-group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* A mother with a child (0-3 years) from the African and/or Caribbean heritage
* Able to provide full consent for their participation
* A resident of the UK
* Able to complete a baseline assessment
* Score 5 or above on Patient Health Questionnaire (PHQ-9)

Exclusion Criteria:

* Less than 18 years
* Medical disorder that would prevent participation in a clinical trial such as Tuberculosis or heart failure
* Temporary residents are unlikely to be available for follow up
* Active suicidal ideation or any other severe mental disorder
* Non-residents of the UK
* Unable to consent
* Patients currently undergoing severe mental health treatment
* Unable to speak the English language fluently
* Other significant physical or learning disability

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in postnatal depression is being assessed | Change is being assessed from baseline, end of intervention, at 3-months and at 6-months post-intervention
  Primary outcome measure would be assessed using the Edinburgh Postnatal Depression Scale
Change in postnatal anxiety is being assessed | Change is being assessed from baseline, end of intervention, at 3-months and at 6-months post-intervention
  Primary outcome measure would be assessed using the Generalised Anxiety Disorder (GAD7) scale
Change in health is being assessed | Change is being assessed from baseline, end of intervention, at 3-months and at 6-months post-intervention
  Primary outcome measure would be assessed using the Patient Health Questionnaire (PHQ-9)
Change in social support is being assessed | Change is being assessed from baseline, end of intervention, at 3-months and at 6-months post-intervention
  Primary outcome measures would be assessed using the Oslo Social Support Scale
Change in health-related quality of life is being assessed | Change is being assessed from baseline, end of intervention, at 3-months and at 6-months post-intervention
  Outcome measure would be assessed using the Health-related Quality of Life scale (EuroQoL-5 Dimensions)
Change in service satisfaction is being assessed | Change is being assessed at end of intervention, at 3-months and at 6-months post-intervention
  Outcome measure would be assessed using the brief Verona Service Satisfaction Scale
Change in child physio-emotional development is being assessed | Change is being assessed from baseline, end of intervention, at 3-months and at 6-months post-intervention
  Outcome measure would be assessed using the Ages and Stages Social-Emotional Questionnaire
Change in parenting knowledge of child development is being assessed | Change is being assessed from baseline, end of intervention, at 3-months and at 6-months post-intervention
  Outcome measure would be assessed using the Learning through Play (LTP) Knowledge, Attitude and Practices (KAP) Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham Trent University, Nottingham, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Jidong DE, Ike TJ, Murshed M, Francis C, Mwankon SB, Jidong JE, Pwajok JY, Nyam PP, Husain N. Postnatal depression in British mothers of African and Caribbean origin: a randomised controlled trial of learning through play plus culturally adapted cognitive behaviour therapy compared with psychoeducation. Front Psychiatry. 2024 Mar 28;15:1383990. doi: 10.3389/fpsyt.2024.1383990. eCollection 2024. PMID 38606412
- [Derived] Jidong DE, Ike JT, Husain N, Murshed M, Francis C, Mwankon BS, Jack BD, Jidong JE, Pwajok YJ, Nyam PP, Kiran T, Bassett P. Culturally adapted psychological intervention for treating maternal depression in British mothers of African and Caribbean origin: A randomized controlled feasibility trial. Clin Psychol Psychother. 2023 May-Jun;30(3):548-565. doi: 10.1002/cpp.2807. Epub 2023 Jan 3. PMID 36478339